CLINICAL TRIAL: NCT00783926
Title: Double Blind, Multi-Center, Phase 1 Study of a Vero Cell-Derived, Whole Virus Clade 2 H5N1 Influenza Vaccine in Healthy Subjects Aged 18 to 45 Years
Brief Title: Phase 1 Study of a H5N1 Influenza Vaccine (Reverse Genetic Reassortant)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alachua Government Services, Inc. (Industry)
Responsible Party: Karen Near, MD; Medical Director, Baxter Healthcare Corporation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 810801
Record Dates: First submitted 2008-10-31; First posted 2008-11-03 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2009-07

CONDITIONS: Influenza; Pandemic Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Experimental): 60 subjects randomized in an equal number to six different vaccine doses
  Interventions: Biological: H5N1 Influenza Vaccine, Whole virion, Vero cell-derived, Inactivated Influenza Vaccine, non-adjuvanted (reverse genetic reassortant/H5N1 hemagglutinin antigen)
- Cohort 2 (Experimental): Following review of safety data of Cohort 1, approximately 360 additional subjects randomized in an equal number to the six different vaccine doses
  Interventions: Biological: H5N1 Influenza Vaccine, Whole virion, Vero cell-derived, Inactivated Influenza Vaccine, non-adjuvanted (reverse genetic reassortant/H5N1 hemagglutinin antigen)

INTERVENTIONS:
Biological: H5N1 Influenza Vaccine, Whole virion, Vero cell-derived, Inactivated Influenza Vaccine, non-adjuvanted (reverse genetic reassortant/H5N1 hemagglutinin antigen) — 2 x 0.5 mL intramuscular injections 21 days apart (one of six different doses of hemagglutinin antigen without adjuvant)

SUMMARY:
The objectives of this study are to assess the dose-related safety and immunogenicity of six different dose levels of inactivated, Vero cell-derived reverse genetic reassortant A/H5N1/Indonesia/05/2005 influenza vaccine in a healthy young adult population. Subjects will receive 2 vaccinations (21 days apart) at the dose to which they were assigned. Blood will be drawn from all subjects for serum antibody determination on Days 0, 21, 42 and 180. Body temperature will be measured daily for 6 days following vaccination. Injection site reactions and systemic reactions will be monitored throughout the entire 180 days of the study. Safety data obtained at 7 days after the first vaccination for all dose levels in Cohort 1 will be reviewed by a Data Monitoring Committee and a recommendation will be obtained whether to proceed to the second vaccination of Cohort 1 and to the first vaccination of Cohort 2.

ELIGIBILITY:
Inclusion Criteria:

Subjects who

* Have an understanding of the study, agree to its provisions, and give written informed consent prior to study entry
* Are clinically healthy, as determined by the Investigator's clinical judgment through collection of medical history and performance of a physical examination
* Are physically and mentally capable of participating in the study
* Are willing to refrain from blood donation for the duration of Part A of the study (until Day 42 [= 21 days after the second vaccination])
* Agree to keep a daily record of symptoms for the duration of the study
* If female and capable of bearing children - have a negative urine pregnancy test result within 24 hours of the scheduled first vaccination and agree to employ adequate birth control measures for the duration of the study.

Exclusion Criteria:

Subjects will be excluded from participation in this study if they:

* Have a history of exposure to H5N1 influenza virus or a history of vaccination with an H5N1 influenza vaccine
* Are at potential occupational risk of contracting H5N1 influenza infection (e.g., poultry workers)
* Suffer from or have a history of a significant neurological, cardiovascular, pulmonary (including asthma), hepatic, rheumatic, autoimmune, hematological, metabolic or renal disorder
* Have a Body Mass Index > 35
* Have hypertension at screening that is graded as greater than Stage 1 (defined as a systolic pressure > 159 or diastolic pressure > 99) while seated and at rest (measurement shall be repeated twice before subject is excluded)
* Have clinically significant abnormal clinical laboratory values at screening as determined by the Investigator
* Have clinically significant electrocardiographic abnormalities at screening
* Test positive for HIV, HBcAb or HCV
* Suffer from any kind of immunodeficiency
* Suffer from a disease or were undergoing a form of treatment within 30 days of study entry or are currently undergoing a form of treatment that can be expected to influence immune response. Such treatment includes, but is not limited to, systemic or high dose inhaled (>800µg/day of beclomethasone dipropionate or equivalent) corticosteroids, radiation treatment or other immunosuppressive or cytotoxic drugs
* Have a history of severe allergic reactions (e.g. clinically severe urticaria, allergic rhinitis, asthma) or anaphylaxis (a medical emergency caused by an acute hypersensitivity reaction involving several organ systems including, but not limited to, cardio-respiratory signs with mucosal and/or skin changes (e.g. angioedema, etc) that presents as or rapidly progresses to a severe life-threatening reaction.
* Have a rash, dermatologic condition or tattoos which may interfere with injection site reaction rating
* Have received any blood products (e.g. a blood transfusion or immunoglobulins within 90 days of vaccination in this study
* Have donated one or more units of blood (approximately 450 mL) or plasma within 30 days of vaccination in this study
* Have received any live vaccine within 4 weeks or an inactivated vaccine or subunit vaccine within 2 weeks prior to vaccination in this study
* Have functional or surgical asplenia
* Have a positive urine drug screen (unless the subject is currently prescribed the drug detected by a licensed health care provider and the continued administration of the drug would not otherwise exclude the subject from participation)
* Have a known or suspected problem with alcohol or drug abuse
* Were administered an investigational drug within six weeks prior to study entry
* Are concurrently participating in a clinical study that includes the administration of an investigational product
* Are a member of the team conducting this study
* Are in a dependent relationship with the study Investigator or with a study team member. Dependent relationships include close relatives (i.e. children, partner/spouse, siblings, parents) as well as employees of the Investigator or site conducting the study
* If female: are pregnant or lactating

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 422 (Actual)
Dates: Start 2008-07; Primary Completion 2009-02 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Number of subjects with an antibody response to the vaccine strain associated with protection 21 days after the second vaccination | 42 days

SECONDARY OUTCOMES:
Frequency and severity of systemic reactions and injection site reactions after the first and second vaccinations | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Baxter BioScience Investigator, MD, Study Director — Baxter Healthcare Corporation
Locations (6):
- United States (6):
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - The Center for Pharmaceutical Research, Kansas City, Missouri
  - Rochester Clinical Research, Rochester, New York
  - Omega Medical Research, Warwick, Rhode Island
  - Research Across America, Dallas, Texas